CLINICAL TRIAL: NCT03777163
Title: Safety and Immunogenicity of the Butantan Institute Trivalent Seasonal Influenza Vaccine in Comparison With the Sanofi Pasteur Trivalent Seasonal Influenza Vaccine in Brazilian Subjects.
Brief Title: Safety and Immunogenicity of the Butantan Institute Influenza Vaccine Compared to Sanofi Pasteur Influenza Vaccine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Butantan Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FLU-07-IB
Record Dates: First submitted 2018-12-12; First posted 2018-12-17 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Influenza
Keywords: Vaccine; Immunization; Safety; Immunogenicity
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Butantan Trivalent Influenza Vaccine (Other): Butantan Institute Trivalent Seasonal Influenza Vaccine (IB-TIV): 15 μg influenza A/H1N1 antigen + 15 μg influenza A/H3N2 antigen + 15 μg influenza B antigen
  Patients will receive one dose (0,5 ml) via intramuscular injection.
  Interventions: Biological: Butantan Institute Trivalent Seasonal Influenza Vaccine
- Sanofi Trivalent Influenza Vaccine (Other): Sanofi Trivalent Seasonal Influenza Vaccine (IB-TIV): 15 μg influenza A/H1N1 antigen + 15 μg influenza A/H3N2 antigen + 15 μg influenza B antigen
  Patients will receive one dose (0,5 ml) via intramuscular injection.
  Interventions: Biological: Sanofi Trivalent Seasonal Influenza Vaccine

INTERVENTIONS:
Biological: Butantan Institute Trivalent Seasonal Influenza Vaccine — Butantan Institute and Pasteur-Mérieux (present, Sanofi Pasteur) established a technology transfer in 1999 for the production of a trivalent influenza vaccine of inactivated split-virion using embryonated eggs. The technology transfer followed a progressive approach from importing the finished product, to packaging and quality control test for release (1999), and, finally, to the first batch of influenza vaccine entirely produced by Butantan (2011). In 2013, the Butantan vaccine was registered by the Brazilian National Agency of Sanitary Surveillance (ANVISA).
  Arms: Butantan Trivalent Influenza Vaccine
Biological: Sanofi Trivalent Seasonal Influenza Vaccine — VAXIGRIP® was launched in 1968 and since then has been licensed in more than 100 countries and prequalified by WHO in 2011. Several clinical studies by Sanofi Pasteur have examined the safety and immunogenicity of Vaxigrip® in older children (8-10 years), adults (18-59 years), elderly (> 60 years),11,12 children (six months to three years) 13 and pregnant women.
  Arms: Sanofi Trivalent Influenza Vaccine

SUMMARY:
The overall aim of this study is to evaluate the safety and immunogenicity of Butantan Institute Trivalent Seasonal Influenza Vaccine in comparison with the Sanofi Trivalent Seasonal Influenza Vaccine.

DETAILED DESCRIPTION:
To detemine whether immunogenicity elicited by a single-dose Butantan Institute Trivalent Seasonal Influenza Vaccine is not inferior to that elicited by a single dose of Sanofi Trivalent Seasonal Influenza Vaccine in adult and elderly populations measured by HI GMT for the three vaccine components 21 days post-immunization.

To describe the safety profile of Butantan Institute Trivalent Seasonal Influenza Vaccine and Sanofi Trivalent Seasonal Influenza Vaccine after a single dose in adult and elderly populations.

ELIGIBILITY:
Inclusion Criteria:

* Adult, male or female, age 18 to 69 years (inclusive) at the time of enrollment;
* Provide written informed consent;
* Agrees to complete all study visits, procedures and contacts;

Exclusion Criteria:

* Chronic medical conditions such as psychiatric conditions, diabetes, hypertension or any other conditions that might place the subjects at high risk of adverse events. Study clinicians will use clinical judgment on a case-by-case basis to assess safety risks under this criterion;
* Clinically significant abnormalities on physical examination;
* Use of immunosuppressive medications such as systemic corticosteroids or chemotherapeutics, or immunosuppressive illness. It will be considered immunosuppressive dose of systemic corticosteroids the equivalent to a dose ≥10 mg of prednisone per day for over 14 days;
* Women who report being pregnant or have plans to become pregnant during the study period;
* Participation in research involving another investigational product within 30 days before planned date of first vaccination or anytime through the last study safety visit;
* Acute febrile illness (axilar temperature ≥ 37.8°C);
* Hypersensitivity to egg or chicken proteins;
* History of Guillain-Barre Syndrome;
* Thrombocytopenia or a bleeding disorder contraindicating intramuscular vaccination;
* Unstable chronic illness (defined as illness requiring hospitalization or a clinically significant change in medication in the previous 12 weeks);
* Alcohol abuse or drug addiction;
* Any vaccination within the previous 4 weeks;
* Seasonal influenza vaccination in the previous 6 months.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 632 (Actual)
Dates: Start 2019-04-22 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Geometric Mean Titers of Hemaglutination Inhibition (HI) for each of the three vaccine components. | 21 days
  HI titers will be determined in serum samples collected before vaccination and 21 days after vaccination from all the subjects.
Adverse events occurring over the immediate 30-minute post vaccination | 30-minute post vaccination
  Immediate Reactogenicity
Number of participants with solicited local AE (erythema, swelling, induration, pain, tenderness, ecchymosis, pruritus) until 3 days post vaccination. | 3 days post vaccination
  Solicited Local Adverse Events
Number of participants with solicited systemic AEs (fever, fatigue, malaise, myalgia, arthralgia, chills, nausea, vomiting, and headache) until 3 days post vaccination. | 3 days post vaccination
  Solicited Systemic Adverse Events
Number of participants with unsolicited adverse events up to 3 days after vaccination. | 3 days after vaccination.
  Unsolicited Adverse Events
All adverse reactions with severity graded 3/4 over the entire study period. | 180 days after vaccination.
  Adverse Reactions with severity graded 3/4

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Precioso, MD, PhD, Study Director — Instituto butantan
Locations (4):
- Brazil (4):
  - Unidade de Pesquisa Clínica do Hospital das Clínicas da Faculdade de Medicina de Ribeirão Preto da Universidade de São Paulo, Ribeirão Preto, São Paulo
  - Centro de Referências para Imunobiológicos Especiais da Universidade Federal de São Paulo, São Paulo, São Paulo
  - Centro de Pesquisas Clínicas do Instituto da Criança do Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo, São Paulo
  - Centro de Referência de Imunobiológicos Especiais (CRIE) Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: No